CLINICAL TRIAL: NCT05692440
Title: Prospective, Single-Arm, Cohort Study on Basivertebral Nerve Ablation With the Intracept Procedure
Brief Title: Basivertebral Nerve Ablation With the Intracept Procedure
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Neuro Spine and Pain Center of Key West (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20223348
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Low Back Pain
Keywords: Basivertebral nerve radiofrequency ablation; Chronic low back pain; Vertebrogenic pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Basivertebral Nerve Ablation (Other): Intraosseous radiofrequency basivertebral nerve ablation
  Interventions: Device: Intracept Procedure

INTERVENTIONS:
Device: Intracept Procedure — Intraosseous radiofrequency ablation of the basivertebral nerve

SUMMARY:
This is an independent prospective, noninterventional, single arm post market data collection of the patient-reported effectiveness, ongoing safety, and satisfaction outcomes for patients treated with intraosseous basivertebral nerve ablation using the Intracept Procedure at a single study site.

DETAILED DESCRIPTION:
Participants in the study will have three study visits over a period of one-year (one prior to procedure and 2 post their procedure). Study visits will be conducted in person by the principal investigator and/or authorized and trained clinical research coordinators at the study site. Participants will be consented and evaluated for inclusion/exclusion criteria and a baseline collect at the initial visit (prior to procedure). Participants will be followed post intraosseous basivertebral nerve ablation at 1, 3, 6, and 12, and 24 months.

Primary and secondary objectives are based on patient reported outcomes for functional improvement (Oswestry Disability Index), low back pain reduction (Visual Analog Scale), and physical and mental health pre and post procedure (EQ-5D-5L and SF-36).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years of age
* Patients who have experienced chronic low back pain for ≥6 months.
* Patients who have not responded to at least 6 months of conservative care.
* Patients with Modic type 1 or 2 changes.

Exclusion Criteria:

* Patients with severe cardiac or pulmonary disease.
* Patients with active systemic infection or localized infection in the treatment area.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-05-03 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) Change- 6 Months | 6 Months
  Validated questionnaire of low back pain related disability. Compromised of 10 questions evaluating the impact of low back pain on activities of daily living. The ODI is scored on a scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). Comparison of mean ODI baseline to 6 months.

SECONDARY OUTCOMES:
Oswestry Disability Index (ODI) Change-12 Months | 12 Months
  Validated questionnaire of low back pain related disability. Comprised of 10 questions evaluating the impact of low back pain on activities of daily living. The ODI is scored on a scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimal disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). Comparison of mean ODI baseline to 6 months. The minimally clinically important difference is a 15-point reduction from baseline.
Visual Analog Scale (VAS)- 6 Months | 6 Months
  Change in the mean visual analog scale (VAS) low back pain score from baseline to 6-months post treatment. VAS in a 10-point numeric scale with a 0 being no pain and 10 being worst imaginable pain. The minimal clinically important difference is a 50% decrease in VAS from baseline.
Visual Analog Scale (VAS)- 12 Months | 12 Months
  Change in the mean visual analog scale (VAS) low back pain score from baseline to 12-months post treatment. VAS is a 10-point numeric scale with 0 being no pain and 10 being worst imaginable pain. The minimally clinically important difference is a 50% decrease in VAS from baseline.
ODI Responder Rate- 6 Months | 6 Months
  Number & percent of patients with greater than or equal to 15-point reduction in Oswestry Disability Index (ODI) from baseline to 6 months post treatment. ODI is scored on a scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimally disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). The minimally clinically important difference is a 15-point reduction from baseline.
ODI Responder Rate- 12 Months | 12 Months
  Number & percent of patients with greater than or equal to 15-point reduction in Oswestry Disability Index (ODI) from baseline to 12 months post treatment. ODI is scored on a scale of 0 (no disability) to 100 (complete disability), with categories of 0-20 (minimally disability), 21-40 (moderate disability), 41-60 (severe disability), 61-80 (crippling back pain), and 81-100 (bed-bound or exaggerating). The minimally clinically important difference is a 15-point reduction from baseline.
VAS Responder Rate- 6 Months | 6 Months
  Number and percentage of participants with a greater than or equal to a 50% reduction from baseline in visual analog scale (VAS) for low back pain at 6 months post treatment. VAS is a patient-reported 10-point numeric pain scale with 0 being no pain and 10 being worst imaginable pain. The minimally clinically important difference in VAS from baseline is a 50% reduction.
VAS Responder Rate-12 Months | 12 Months
  Number and percentage of participants with a greater than or equal to a 50% reduction from baseline in visual analog scale (VAS) for low back pain at 12 months post treatment. VAS is a patient-reported 10-point numeric pain scale with 0 being no pain and 10 being worst imaginable pain. The minimal clinically important difference in VAS from baseline is a 50% reduction.

CONTACTS AND LOCATIONS:
Overall Officials: William Schnapp, PhD, Principal Investigator — Owner
Locations (1):
- Neuro Spine and Pain Center of Key West, Key West, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schnapp W, Schnapp M, Gottlieb J, Alexandre LC, Martiatu K, Delcroix GJ. Prospective cohort study of basivertebral nerve ablation for chronic low back pain in a real-world setting: 12 months follow-up. Interv Pain Med. 2024 Nov 25;3(4):100446. doi: 10.1016/j.inpm.2024.100446. eCollection 2024 Dec. PMID 39655088